CLINICAL TRIAL: NCT01109992
Title: Integrated Dual Exercise and Lexiscan PET: IDEAL PET
Brief Title: Integrated Dual Exercise and Lexiscan Positron Emission Tomography: IDEALPET
Acronym: IDEALPET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sharmila Dorbala, MBBS, Director, Nuclear Cardiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BWH
Record Dates: First submitted 2010-04-16; First posted 2010-04-23 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; exercise; regadenoson; positron emission tomography
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity | interventions — Exercise; regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regadenoson (Lexiscan) (Active Comparator): Regadenoson Rubidium-82 Positron Emission Tomography
  Interventions: Drug: Regadenoson (Lexiscan)
- Exercise + Regadenoson (Lexercise) (Experimental): Exercise plus Regadenoson (Lexercise) Rubidium-82 Positron Emission Tomography
  Interventions: Drug: Exercise plus Regadenoson (Lexercise)

INTERVENTIONS:
Drug: Exercise plus Regadenoson (Lexercise) — Standard Bruce exercise stress test with regadenoson injection at maximal stress with Rubidium-82 Positron Emission Tomography
  Other Names: Exercise plus Lexiscan
  Arms: Exercise + Regadenoson (Lexercise)
Drug: Regadenoson (Lexiscan) — Regadenoson Rubidium-82 Positron Emission Tomography
  Arms: Regadenoson (Lexiscan)

SUMMARY:
This is a single-center study of subjects undergoing clinically indicated heart scans for evaluation of known or suspected heart disease. We will also include 10 healthy subjects without known heart disease. We would like to study stress testing of the heart using exercise and a medication called regadenoson. Imaging of the heart will be performed.

DETAILED DESCRIPTION:
Regadenoson is stress agent approved by the FDA for use with myocardial perfusion imaging with technetium-99m single photon emission computed tomography (SPECT) in patients that are unable to exercise adequately. We would like to study Regadenoson in conjunction with Exercise Rubidium-82 positron emission tomography myocardial perfusion imaging (PET MPI). Regadenoson is not approved by FDA for use with Rubidium-82 PET MPI. Also, we would like to study a novel stress protocol of Regadenoson combined with symptom limited exercise stress (not FDA approved).

The objectives of this study are to assess the tolerability and safety of combined symptom limited exercise stress test with Lexiscan (Lexercise PET) compared to Lexiscan alone (Lexiscan PET), to assess image quality of Lexercise compared to Lexiscan PET and to compare relative and absolute myocardial perfusion imaging with Lexercise compared to Lexiscan PET to identify CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinically indicated N-13 ammonia PET study or ten healthy volunteers
* Known coronary artery disease (prior percutaneous coronary intervention, prior coronary artery bypass surgery or Q wave MI on ECG) or intermediate to high pretest likelihood of CAD
* Able to exercise on a treadmill
* Able and willing to provide informed consent to participate in the study

Exclusion Criteria:

* Contraindications to exercise stress testing such as, unstable angina, known severe left main coronary artery stenosis, severe heart failure, uncontrolled arrhythmias, symptomatic hypotension or severe hypertension (systolic blood pressure < 90 or > 200 mmHg, respectively), or > 1st degree atrioventricular block in the absence of a functioning pacemaker.
* Subject requires emergent cardiac medical intervention or catheterization after the clinical study.
* Documented myocardial infarction (MI) ≤ 30 days prior to enrollment.
* History of percutaneous coronary intervention (PCI) ≤ 4weeks prior to enrollment.
* History of coronary artery bypass graft (CABG) ≤ 8 weeks prior to enrollment.
* History of heart transplantation.
* Allergy or intolerance to aminophylline or regadenoson
* Known severe or oxygen dependent bronchoconstrictive or bronchospastic lung disease [e.g., asthma, wheezing, chronic obstructive pulmonary disease (COPD), etc.].
* Severe LV dysfunction, with ejection fraction of < 30%
* Serious non-cardiac medical illness (e.g., disseminated malignancy, severe neurological dysfunction at time of baseline PET study) or a social situation which will preclude research study participation
* History of Seizures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Dorbala, MBBS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Womens' Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Chow BJ, Ananthasubramaniam K, dekemp RA, Dalipaj MM, Beanlands RS, Ruddy TD. Comparison of treadmill exercise versus dipyridamole stress with myocardial perfusion imaging using rubidium-82 positron emission tomography. J Am Coll Cardiol. 2005 Apr 19;45(8):1227-34. doi: 10.1016/j.jacc.2005.01.016. PMID 15837254
- [Background] Di Carli MF, Hachamovitch R. New technology for noninvasive evaluation of coronary artery disease. Circulation. 2007 Mar 20;115(11):1464-80. doi: 10.1161/CIRCULATIONAHA.106.629808. No abstract available. PMID 17372188
- [Background] Klocke FJ, Baird MG, Lorell BH, Bateman TM, Messer JV, Berman DS, O'Gara PT, Carabello BA, Russell RO Jr, Cerqueira MD, St John Sutton MG, DeMaria AN, Udelson JE, Kennedy JW, Verani MS, Williams KA, Antman EM, Smith SC Jr, Alpert JS, Gregoratos G, Anderson JL, Hiratzka LF, Faxon DP, Hunt SA, Fuster V, Jacobs AK, Gibbons RJ, Russell RO; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American Society for Nuclear Cardiology. ACC/AHA/ASNC guidelines for the clinical use of cardiac radionuclide imaging--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/ASNC Committee to Revise the 1995 Guidelines for the Clinical Use of Cardiac Radionuclide Imaging). Circulation. 2003 Sep 16;108(11):1404-18. doi: 10.1161/01.CIR.0000080946.42225.4D. No abstract available. PMID 12975245
- [Background] Chow BJ, Beanlands RS, Lee A, DaSilva JN, deKemp RA, Alkahtani A, Ruddy TD. Treadmill exercise produces larger perfusion defects than dipyridamole stress N-13 ammonia positron emission tomography. J Am Coll Cardiol. 2006 Jan 17;47(2):411-6. doi: 10.1016/j.jacc.2005.09.027. PMID 16412870
- [Background] Camici PG, Crea F. Coronary microvascular dysfunction. N Engl J Med. 2007 Feb 22;356(8):830-40. doi: 10.1056/NEJMra061889. No abstract available. PMID 17314342
- [Background] El Fakhri G, Sitek A, Guerin B, Kijewski MF, Di Carli MF, Moore SC. Quantitative dynamic cardiac 82Rb PET using generalized factor and compartment analyses. J Nucl Med. 2005 Aug;46(8):1264-71. PMID 16085581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 subjects consented for the study and 41 subjects completed the study. One subject did not come for the study procedures. One subject could not cooperate with imaging and was moving during the rest scan. Regadenoson scan was not performed.
Groups:
- Regadenoson: Regadenoson Rubidium-82 Positron Emission Tomography
  Regadenoson Rubidium-82 Positron Emission Tomography
- Exercise + Regadenoson: Exercise plus Regadenoson Rubidium-82 Positron Emission Tomography
  Exercise plus Regadenoson: Standard Bruce exercise stress test with regadenoson injection at maximal stress with Rubidium-82 Positron Emission Tomography
Period: Overall Study
Arm/Group | Regadenoson | Exercise + Regadenoson
Started (Subjects screened) | 11 | 32
Subjects Enrolled | 11 | 32
Completed | 11 | 30
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Movement during rest scan. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Regadenoson: Regadenoson Rubidium-82 Positron Emission Tomography
  Regadenoson: Regadenoson Rubidium-82 Positron Emission Tomography
- Total: Total of all reporting groups
Arm/Group | Regadenoson | Exercise + Regadenoson | Total
Number analyzed (Participants) | 11 | 30 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11) | 54 (15) | 57 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 14 | 17
  Male | 8 | 16 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 9 | 22 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 30 | 41

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Combined Exercise and Regadenoson Stress
Description: 1. Count of subjects with ischemic ECG changes is reported
  2. Count of subjects with systolic blood pressure decrease > 20 mm Hg is reported
  3. Count of subjects with abnormal serum troponin T levels is reported
  4. Radiation dose to the staff will be measured using personal dosimeters after the Lexiscan as well as the Lexercise PET study.
Time Frame: Day of the research scan during the stress test
Population: Radiation dose to staff was not measured due to logistical difficulties.Three subjects had blood pressure changes in the Regadenoson (Lexiscan) arm; 3 subjects showed ischemic ECG changes in the exercise + regadenoson (Lexercise) arm; and, none of the subjects showed abnormal troponin levels.
Measure: Count of Participants; unit: Participants
Arm/Group | Regadenoson (Lexiscan) | Exercise + Regadenoson (Lexercise)
Number analyzed (Participants) | 11 | 30
Participants
  Count of ischemic ECG changes | 0 | 3
  Count of subjects systolic blood pressure decrease | 3 | 0
  Count of subjects with abnormal troponin | 0 | 0

2. Secondary Outcome: Image Quality: Heart to Liver Ratio of Counts
Description: Sub-diaphragmatic activity: Heart to Liver Ratio was measured on the rubidium-82 and N-13 ammonia scans. Since this measure is a ratio it has no units. Mean and Standard Deviation of Ratio is reported for each group.
  This was measured on the clinical scan and on the research scan which were performed about 2 weeks apart in most subjects.
Time Frame: Week 1 (day of the clinical scan), and Week 2 (day of the research scan)
Measure: Mean (Standard Deviation); unit: mean ratio
Groups:
- Regadenoson (Lexiscan): Regadenoson Rubidium-82 Positron Emission Tomography
  Regadenoson (Lexiscan): Regadenoson Rubidium-82 Positron Emission Tomography.
  No adverse events
- Exercise + Regadenoson (Lexiscan): Exercise plus Regadenoson (Lexiscan) Rubidium-82 Positron Emission Tomography
  Exercise plus Regadenoson (Lexercise): Standard Bruce exercise stress test with regadenoson injection at maximal stress with Rubidium-82 Positron Emission Tomography
  No adverse events
Arm/Group | Regadenoson (Lexiscan) | Exercise + Regadenoson (Lexiscan)
Number analyzed (Participants) | 11 | 30
mean ratio
  Stress Scan 1 | 1.23 (0.55) | 1.11 (0.58)
  Stress Scan 2 | 1.25 (0.57) | 1.37 (0.82)

3. Secondary Outcome: Changes in Left Ventricular Function With Dual Exercise and Regadenoson PET
Description: Left ventricular ejection fraction (LVEF) at stress was measured at Stress scan 1 (regadenoson) and Stress scan 2 (regadenoson or exercise + regadenoson).
  This was measured on the clinical scan and on the research scan which were performed about 2 weeks apart in most subjects.
Time Frame: Week 1 (day of the clinical scan), and Week 2 (day of the research scan)
Measure: Mean (Standard Deviation); unit: percentage of LVEF
Groups:
- Exercise + Regadenoson (Lexercise): Exercise plus Regadenoson (Lexercise) Rubidium-82 Positron Emission Tomography
  Exercise plus Regadenoson (Lexercise): Standard Bruce exercise stress test with regadenoson injection at maximal stress with Rubidium-82 Positron Emission Tomography
  No adverse events
Arm/Group | Regadenoson (Lexiscan) | Exercise + Regadenoson (Lexercise)
Number analyzed (Participants) | 11 | 30
percentage of LVEF
  Stress 1 Scan | 58 (15) | 60 (14)
  Stress 2 Scan | 59 (15) | 62 (14)

4. Secondary Outcome: Peak Stress Myocardial Blood Flow
Description: Myocardial Blood Flow Measured at Peak Hyperemia With Regadenoson or Immediately After Exercise + Regadenoson This was measured on the clinical scan and on the research scan which were performed about 2 weeks apart in most subjects.
Time Frame: Week 1 (day of the clinical scan), and Week 2 (day of the research scan)
Population: Myocardial blood flow could not be accurately measured in one subject from each arm. Therefore we report information on 10/11 subjects in Regadenoson arm and 29/30 subjects in the Exercise + Regadenoson arm.
Measure: Mean (Standard Deviation); unit: mL/gm/min
Arm/Group | Regadenoson (Lexiscan) | Exercise + Regadenoson (Lexiscan)
Number analyzed (Participants) | 10 | 29
mL/gm/min
  Stress 1 Scan | 1.82 (0.73) | 2.04 (0.58)
  Stress 2 Scan | 1.85 (0.85) | 2.34 (0.82)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on the day of the research study which was in week 2 for most patients.
Groups:
- Exercise + Regadenoson (Lexiscan): Exercise plus Regadenoson (Lexiscan) Rubidium-82 Positron Emission Tomography
  Exercise plus Regadenoson (Lexercise): Standard Bruce exercise stress test with regadenoson injection at maximal stress with Rubidium-82 Positron Emission Tomography
Arm/Group | Regadenoson (Lexiscan) | Exercise + Regadenoson (Lexiscan)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/30
Other Adverse Events (participants affected / at risk) | 0/11 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT01109992/Prot_SAP_000.pdf